CLINICAL TRIAL: NCT02478918
Title: Automated Telephone Reminder Prior to Outpatient Colonoscopy and the Effect on Bowel Preparation Quality
Brief Title: Automated Telephone Reminder for Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Lawrence Hookey, MD, Division of Gastroenterology, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 6013364
Record Dates: First submitted 2015-06-18; First posted 2015-06-23 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Polyps
MeSH Terms: conditions — Polyps

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Receiving reminder phone call (Experimental): Will receive phone call to remind colonoscopy date and bowel prep
  Interventions: Other: Phone call
- Not receiving reminder phone call (No Intervention): Will not receive phone call to remind colonoscopy date and bowel prep

INTERVENTIONS:
Other: Phone call — Automated phone call reminder
  Arms: Receiving reminder phone call

SUMMARY:
This is a quality improvement study to determine the impact of an automated telephone reminder on the quality of bowel preparation in patients undergoing outpatient colonoscopy.

DETAILED DESCRIPTION:
Randomized trial of automated reminders with bowel prep instructions and encouraging clear fluid ingestion. The phone calls will occur 48-96 hours prior to the scheduled colonoscopy.

All patients undergoing outpatient colonoscopy and prescribed sodium picosulfate plus magnesium citrate will be eligible for enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Scheduled for outpatient colonoscopy at a later date
* Prescribed evening-before or split-dose low volume preparation regimens

Exclusion Criteria:

* Refusal to receive automated telephone reminder
* No access to telephone
* Urgent/emergent indication for colonoscopy
* Prescribed a bowel prep other than Pico-Salax/Purgodan
* Receiving upper and lower combined procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2015-06; Primary Completion 2016-05-15 (Actual); Study Completion 2016-05-15 (Actual)

PRIMARY OUTCOMES:
Ottawa preparation scale score | Immediately after procedure
  measures the cleanliness of each part of the colon and the overall fluid volume as assessed by the endoscopist

SECONDARY OUTCOMES:
Number of glasses of fluid consumed pre-colonoscopy | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Hookey, MD, Principal Investigator — Queen's University; Matthew Church, Study Director — Queen's University; Natalie Rubinger, Study Director — Queen's University
Locations (1):
- Hotel Dieu Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abuksis G, Mor M, Segal N, Shemesh I, Morad I, Plaut S, Weiss E, Sulkes J, Fraser G, Niv Y. A patient education program is cost-effective for preventing failure of endoscopic procedures in a gastroenterology department. Am J Gastroenterol. 2001 Jun;96(6):1786-90. doi: 10.1111/j.1572-0241.2001.03872.x. PMID 11419830
- [Background] Calderwood AH, Lai EJ, Fix OK, Jacobson BC. An endoscopist-blinded, randomized, controlled trial of a simple visual aid to improve bowel preparation for screening colonoscopy. Gastrointest Endosc. 2011 Feb;73(2):307-14. doi: 10.1016/j.gie.2010.10.013. Epub 2010 Dec 18. PMID 21168840
- [Background] Liu X, Luo H, Zhang L, Leung FW, Liu Z, Wang X, Huang R, Hui N, Wu K, Fan D, Pan Y, Guo X. Telephone-based re-education on the day before colonoscopy improves the quality of bowel preparation and the polyp detection rate: a prospective, colonoscopist-blinded, randomised, controlled study. Gut. 2014 Jan;63(1):125-30. doi: 10.1136/gutjnl-2012-304292. Epub 2013 Mar 16. PMID 23503044
- [Background] Modi C, Depasquale JR, Digiacomo WS, Malinowski JE, Engelhardt K, Shaikh SN, Kothari ST, Kottam R, Shakov R, Maksoud C, Baddoura WJ, Spira RS. Impact of patient education on quality of bowel preparation in outpatient colonoscopies. Qual Prim Care. 2009;17(6):397-404. PMID 20051190
- [Background] Ness RM, Manam R, Hoen H, Chalasani N. Predictors of inadequate bowel preparation for colonoscopy. Am J Gastroenterol. 2001 Jun;96(6):1797-802. doi: 10.1111/j.1572-0241.2001.03874.x. PMID 11419832
- [Background] Rostom A, Jolicoeur E. Validation of a new scale for the assessment of bowel preparation quality. Gastrointest Endosc. 2004 Apr;59(4):482-6. doi: 10.1016/s0016-5107(03)02875-x. PMID 15044882
- [Background] Shaikh AA, Hussain SM, Rahn S, Desilets DJ. Effect of an educational pamphlet on colon cancer screening: a randomized, prospective trial. Eur J Gastroenterol Hepatol. 2010 Apr;22(4):444-9. doi: 10.1097/MEG.0b013e328333fca6. PMID 19940781
- [Background] Shieh TY, Chen MJ, Chang CW, Hung CY, Hu KC, Kuo YC, Shih SC, Wang HY. Effect of physician-delivered patient education on the quality of bowel preparation for screening colonoscopy. Gastroenterol Res Pract. 2013;2013:570180. doi: 10.1155/2013/570180. Epub 2013 Dec 17. PMID 24454341
- [Background] Spiegel BM, Talley J, Shekelle P, Agarwal N, Snyder B, Bolus R, Kurzbard N, Chan M, Ho A, Kaneshiro M, Cordasco K, Cohen H. Development and validation of a novel patient educational booklet to enhance colonoscopy preparation. Am J Gastroenterol. 2011 May;106(5):875-83. doi: 10.1038/ajg.2011.75. Epub 2011 Apr 12. PMID 21483463
- [Background] Tae JW, Lee JC, Hong SJ, Han JP, Lee YH, Chung JH, Yoon HG, Ko BM, Cho JY, Lee JS, Lee MS. Impact of patient education with cartoon visual aids on the quality of bowel preparation for colonoscopy. Gastrointest Endosc. 2012 Oct;76(4):804-11. doi: 10.1016/j.gie.2012.05.026. Epub 2012 Jul 27. PMID 22840295